CLINICAL TRIAL: NCT03529903
Title: MyLife: A Digital Health Coaching Program Encouraging Healthy Behaviors in Patients at Risk for Lifestyle-related Chronic Diseases
Brief Title: MyLife: A Digital Health Coaching Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel M. Croymans, MD, MBA, MS, Co-Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-000325
Record Dates: First submitted 2018-04-20; First posted 2018-05-18 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Lifestyle-related Condition; Obesity; Sedentary Lifestyle; PreDiabetes; Hypertension
Keywords: behavior change; health coaching; wearable activity tracker; text messaging; lifestyle-related chronic diseases
MeSH Terms: conditions — Mental Disorders; Obesity; Sedentary Behavior; Prediabetic State; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): *Complete an online survey and intake appointment with a trained Health Coach (HC), who will measure their height, weight, and blood pressure, assess their current health habits (sleep, nutrition, exercise) and work with they to set realistic, achievable health goals. *Wear a Fitbit device daily to track physical activity and weight (members of the MyLife study team can access their data during throughout the program and de-identified, anonymous, data will be shared with Fitbit as part of a research partnership). *Complete another online survey and telephone check-in with their HC at the halfway point to monitor their progress toward reaching their goals. *Complete a final online survey and outtake appointment with their HC to re-check their measurements and discuss their progress.
- Experimental Group (Experimental): *Complete survey/ intake appointment with a HC, who will measure their height, weight, and blood pressure, assess their health habits and set achievable health goals. *Wear a Fitbit to track their daily physical activity and weight *Set a weekly active minutes goal and record their weight weekly. *Receive motivational text messages 4x per week, one will ask for their weekly active minutes goal and weight and another will ask for goal progression.*Complete photo food diaries biweekly (send pictures of everything they eat/drink to their HC). *Complete surveys/telephone check-ins with their HC every 2 weeks to monitor their progress toward reaching their goals. *Complete final survey/outtake appointment with their HC to for final measurements and to discuss goal progression (about 2 hours).
  Interventions: Behavioral: Health Coaching

INTERVENTIONS:
Behavioral: Health Coaching — Our trained health coaches will use the Way To Health platform to track patient health behaviors, and will communicate with patients via both SMS text messaging (up to four messages per week) and biweekly phone calls (up to one hour). During these interactions, health coaches will connect the patient to helpful resources and to help them reflect on previous goals and to set realistic, achievable goals for the upcoming weeks.
  Arms: Experimental Group

SUMMARY:
Lifestyle behaviors such as sleep, diet, and physical activity, are implicated in a number of chronic conditions including hypertension, obesity, diabetes, heart failure, and obstructive sleep apnea. Research shows that despite awareness of this fact, patients at risk for lifestyle-related chronic diseases have difficulty adhering to lifestyle change recommendations made by their physicians, and face challenges when attempting to modify unhealthy behaviors. New technologies, such as wearable activity trackers and automated text messaging, are promising tools for monitoring and promoting healthy lifestyle behaviors among patients. This randomized controlled trial will evaluate the effect of a digital health program, which uses pre-medical post-baccalaureate or undergraduate health coaches, wearable activity trackers (Fitbit Charge 2), and mobile messaging, compared to wearable activity trackers (Fitbit Charge 2) alone in promoting lifestyle change among overweight and sedentary 18-64 year old patients recruited from UCLA Health primary care clinics.

DETAILED DESCRIPTION:
100 overweight and sedentary patients at early risk for lifestyle-related chronic diseases will be recruited and receive a screening and consent survey link via the Way To Health web portal, https://www.waytohealth.org/. Upon reaching the portal, potential participants will be asked to create an account and will then be informed of the details of the study, including its objectives, duration, requirements, and financial payments. If participants are still interested in participating, the Way to Health portal will take them through an automated online informed consent. The consent document will be divided into sections and potential participants will have to click a button to advance through each section. This is to help ensure that participants read the consent form thoroughly by breaking down the form into manageable blocks of text. Successive screens will explain the voluntary nature of the study, the risks and benefits of participation, alternatives to participation, and that participants can withdraw from the study at any time. On the final consent screen, potential participants who click a clearly delineated button stating that they agree to participate in the study will be considered to have consented to enroll. After consenting, participants will complete an online questionnaire to determine their eligibility. Eligible participants will then be randomized using a computer-generated simple randomization algorithm to allocate patients equally (1:1) to one of the study arms (intervention and control) and will be directed to sign up for their intake clinic visit via an online scheduling site. Participants will be provided with details regarding how to contact the research team via email or phone at any time if they subsequently wish to withdraw from the study. This contact information will remain easily accessible via the participants' individual Way to Health web portal dashboards throughout the study. Both health coaches and patients will have portals on the Way To Health platform, in which surveys will be developed and completed. Health coaches will be able to use this portal to track patient progress, including Fitbit physical activity data, while patients will be able to upload pictures (and messages if they choose). Additionally, both automated and manual branching logic text messages will be sent by health coaches via this platform, while patients can respond without using the online application.

Patients will also be required to enter their credit card or debit card information into a secure online service, which will be to apply fees for failure to participate in the study, a total maximum of $150. This information includes the full name associated with the card, complete card number, expiration date, security code/CVV, and billing ZIP code. All patients will be sent multiple participation reminders via email, text message, and phone call. However, patients who ultimately fail to participate in the midpoint survey (approximately 8 weeks in the study) or the outtake survey and associated outtake visit (approximately 16 weeks in the study) will be charged $75 or $75, respectively. Patients who complete the midpoint survey, outtake survey, and outtake clinic visit will be charged $0. All participants will be able to keep their device after the 16 week program is finished. This financial incentive leverages the concept of loss aversion, that "losses loom larger than gains" (Kahneman & Tversky, 1979), to motivate study enrollment and completion rates independent of study arm. Patients may be reimbursed any charge should we receive a note from their primary care physician justifying a medical reason for failure to participate. In addition, if at the end of the study the patient states that they are unable to meet the financial requirement, they will be given the option to return a functional Fitbit for a full reimbursement.

At their intake appointment, patients will meet with study personnel, who will measure their baseline height, weight, and blood pressure. Participants will then complete an intake survey that will assess their lifestyle habits in three areas: sleep, physical activity, and diet/nutrition. The surveys will also assess their personal engagement in their health and baseline level of stress. Based on the responses to these questions, participants in the intervention arm will be assigned a personal health coach and receive health behavior counseling as well as an individualized lifestyle plan, including recommendations and patient-defined goals in each of the three areas. All patients enrolled into the study will receive a free Fitbit™ Charge 2 device during their intake visit appointment (face value of $150) and will be informed of the CDC/federal recommendation guidelines for physical activity (https://www.cdc.gov/physicalactivity/index.html) and nutrition (https://health.gov/dietaryguidelines/2015/guidelines/executive-summary/). Their device will remain free as long as they complete the intake and outtake clinic appointments and complete their intake, midpoint, and outtake surveys (approximate time commitment of 6 hours).

In the intervention group patients will be asked to:

Complete an online survey and intake appointment (about 2 hours) with a trained Health Coach, who will measure their height, weight, and blood pressure, assess their current health habits (sleep, nutrition, exercise) and work with them to set realistic, achievable health goals Wear and use a wearable Fitbit device every day to track their minutes of physical activity and weight (members of the MyLife study team can access their data during throughout the program and de-identified, anonymous, data will be shared with Fitbit as part of a research partnership) Set a weekly active minutes goal and record their weight every week Receive motivational text messages four times per week, including one asking for their weekly active minutes goal and weight and another asking for their progress toward that goal Complete photo food diaries every 2 weeks in which they send pictures of everything they eat or drink to their Health Coach Complete online surveys and telephone check-ins with their Health Coach (about 1 hour total) every 2 weeks to monitor their progress toward reaching their goals Complete a wrap-up online survey and outtake appointment with their Health Coach to re-check their measurements and discuss their progress (about 2 hours)

If they are in the control group patients will be asked to:

Complete an online survey and intake appointment (about 2 hours) with a trained Health Coach, who will measure their height, weight, and blood pressure, assess their current health habits (sleep, nutrition, exercise) and work with they to set realistic, achievable health goals Wear and use a wearable Fitbit device every day to track their minutes of physical activity and weight (members of the MyLife study team can access their data during throughout the program and de-identified, anonymous, data will be shared with Fitbit as part of a research partnership) Complete another online survey and telephone check-in with their Health Coach (about 1 hour total) at the halfway point to monitor their progress toward reaching their goals Complete a wrap-up online survey and outtake appointment with their Health Coach to re-check their measurements and discuss their progress (about 2 hours)

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* English speaking
* Owns a smartphone with texting capabilities.
* BMI >= 27
* Desire to lose weight and increase physical activity.
* Sedentary behavior (defined as less than 150 minutes per week of moderate to vigorous physical activity (MVPA)).
* Have a UCLA Health Primary Care Physician (PCP) and their PCP's agreement to enroll in the study.

Exclusion Criteria:

* Age <18 or > 65
* Does not own a smart-phone
* Currently using a wearable device that tracks physical activity and sleep
* Poorly controlled diabetes mellitus, defined by, but not limited to: o Most recent HbA1c >9 o Diabetic neuropathy that has led to osteomyelitis and/or amputation
* Chronic kidney disease (CKD) grade III or higher OR dialysis dependent
* Chronic heart failure (CHF) stage II or higher
* Unable to participate in physical activity due to chronic medical condition, including, but not limited to: o Severe/advanced joint arthritis o Unstable angina o History of NSTEMI (non-ST elevation myocardial infarction), STEMI (ST elevation myocardial infarction) or stroke in past 12 months oActive cancer undergoing chemotherapy or radiation oActive substance abuse or alcoholism
* Current participation in organized exercise program on a regular or repeated basis defined as coaching sessions at a frequency greater than 4 times per month (ie- Weight Watchers, personalized coaching for nutrition/personal training, and/or cardiac or stroke rehab)
* Any health condition that would limit life expectancy to less than 1 year
* Any additional health condition including cognitive dysfunction, mental health, or physical condition that would prevent patient from participating fully in activity and/or health coaching as defined by their primary care provider (PCP).
* Currently enrolled in any research studies that may influence your physical activity, food and beverage choices, or bodyweight
* Lost more than 10 lbs in the last 3 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Weight | 16 weeks (measured biweekly)
  Weight measured using a scale
Change in Physical Activity | 16 weeks (measured biweekly)
  Activity minutes measured using a wearable activity tracker

CONTACTS AND LOCATIONS:
Overall Officials: Alice Kuo, MD, PhD, MBA, Principal Investigator — Chief of Medicine-Pediatrics, UCLA Health; Daniel M Croymans, MD, MBA, MS, Principal Investigator — Department of Medicine, UCLA Health; Paul J Bixenstine, MD, Principal Investigator — Department of Medicine and Department of Pediatrics, UCLA Health
Locations (1):
- UCLA Medicine - Pediatrics Comprehensive Care Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Dusseldorp E, van Genugten L, van Buuren S, Verheijden MW, van Empelen P. Combinations of techniques that effectively change health behavior: evidence from Meta-CART analysis. Health Psychol. 2014 Dec;33(12):1530-40. doi: 10.1037/hea0000018. Epub 2013 Nov 25. PMID 24274802
- [Background] Patel MS, Asch DA, Volpp KG. Wearable devices as facilitators, not drivers, of health behavior change. JAMA. 2015 Feb 3;313(5):459-60. doi: 10.1001/jama.2014.14781. No abstract available. PMID 25569175
- [Background] Godino JG, Merchant G, Norman GJ, Donohue MC, Marshall SJ, Fowler JH, Calfas KJ, Huang JS, Rock CL, Griswold WG, Gupta A, Raab F, Fogg BJ, Robinson TN, Patrick K. Using social and mobile tools for weight loss in overweight and obese young adults (Project SMART): a 2 year, parallel-group, randomised, controlled trial. Lancet Diabetes Endocrinol. 2016 Sep;4(9):747-755. doi: 10.1016/S2213-8587(16)30105-X. Epub 2016 Jul 14. PMID 27426247
- [Background] Mishuris RG, Yoder J, Wilson D, Mann D. Integrating data from an online diabetes prevention program into an electronic health record and clinical workflow, a design phase usability study. BMC Med Inform Decis Mak. 2016 Jul 11;16:88. doi: 10.1186/s12911-016-0328-x. PMID 27401606
- [Background] Goldman ML, Ghorob A, Eyre SL, Bodenheimer T. How do peer coaches improve diabetes care for low-income patients?: a qualitative analysis. Diabetes Educ. 2013 Nov-Dec;39(6):800-10. doi: 10.1177/0145721713505779. Epub 2013 Oct 29. PMID 24168838